CLINICAL TRIAL: NCT02480712
Title: A Phase 3, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks in Subjects With Chronic Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV)-1 Coinfection
Brief Title: Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Adults With Chronic Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV)-1 Coinfection
Acronym: ASTRAL-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1202
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL (Experimental): Participants will receive SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) for 12 weeks in participants with chronic HCV infection who were coinfected with HIV-1.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV RNA ≥ 10^4 IU/mL at screening
* HCV genotype 1, 2, 3, 4, 5, 6
* Cirrhosis determination, a fibroscan or liver biopsy may be required
* HIV-1 infection
* Use of protocol specified method(s) of contraception
* Screening laboratory values within defined thresholds

Key Exclusion Criteria:

* Clinically-significant illness (other than HCV or HIV) or any other major medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol
* Current or prior history of clinical hepatic decompensation, hepatocellular carcinoma (HCC) or other malignancy (with the exception of certain resolved skin cancers)
* Screening ECG with clinically significant abnormalities
* Pregnant or nursing female or male with pregnant female partner
* Infection with hepatitis B virus (HBV)
* Use of any prohibited concomitant medications as described in the protocol
* Chronic use of systemically administered immunosuppressive agents

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- United States (15):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Wyles D, Brau N, Kottilil S, Daar E, Workowski K, Luetkemeyer A, et al. Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Patients Co-Infected with HCV and HIV-1: The Phase 3 ASTRAL-5 Study [Abstract PS104]. 2016 European Association for the Study of the Liver (EASL), Barcelona, Spain.
- [Derived] Wyles D, Brau N, Kottilil S, Daar ES, Ruane P, Workowski K, Luetkemeyer A, Adeyemi O, Kim AY, Doehle B, Huang KC, Mogalian E, Osinusi A, McNally J, Brainard DM, McHutchison JG, Naggie S, Sulkowski M; ASTRAL-5 Investigators. Sofosbuvir and Velpatasvir for the Treatment of Hepatitis C Virus in Patients Coinfected With Human Immunodeficiency Virus Type 1: An Open-Label, Phase 3 Study. Clin Infect Dis. 2017 Jul 1;65(1):6-12. doi: 10.1093/cid/cix260. PMID 28369210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 17 study sites in the United States. The first participant was screened on 01 July 2015. The last study visit occurred on 22 June 2016.
Pre-assignment Details: 149 participants were screened.
Groups:
- SOF/VEL 12 Weeks: Sofosbuvir/velpatasvir (SOF/VEL; Epclusa®) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1
Period: Overall Study
Arm/Group | SOF/VEL 12 Weeks
Started | 107
Completed | 96
Not Completed | 11
Not completed — Enrolled but Never Treated | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrew Consent | 3
Not completed — Death | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who received at least one dose of study drug.
Groups:
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 48
  White | 54
  Asian | 3
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 91
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 24
    CT | 52
    TT | 30
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.3 (0.57)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 28
  ≥ 800,000 IU/mL | 78
HIV RNA category [Count of Participants; unit: Participants] — Population: Participants in the Safety Analysis Set were analyzed by tenofovir disoproxil fumarate(TDF)-containing antiretroviral therapy (ART) at baseline:
  * Boosted TDF-containing regimens
  * Non-boosted TDF-containing regimens
  * Non TDF-containing regimens
  Participants
    Boosted TDF Containing Regimens: number analyzed (Participants) | 56
    Boosted TDF Containing Regimens: HIV RNA < 50 copies/mL | 55
    Boosted TDF Containing Regimens: HIV RNA ≥ 50 copies/mL | 1
    Non-Boosted TDF Containing Regimens: number analyzed (Participants) | 35
    Non-Boosted TDF Containing Regimens: HIV RNA < 50 copies/mL | 35
    Non-Boosted TDF Containing Regimens: HIV RNA ≥ 50 copies/mL | 0
    Non TDF Containing Regimens: number analyzed (Participants) | 15
    Non TDF Containing Regimens: HIV RNA < 50 copies/mL | 14
    Non TDF Containing Regimens: HIV RNA ≥ 50 copies/mL | 1
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] — Population: Participants in the Safety Analysis Set were analyzed by TDF-containing ART at baseline:
  * Boosted TDF-containing regimens
  * Non-boosted TDF-containing regimens
  * Non TDF-containing regimens
  mg/dL
    Boosted TDF Containing Regimens: number analyzed (Participants) | 56
    Boosted TDF Containing Regimens | 1.02 (0.194)
    Non-Boosted TDF Containing Regimens: number analyzed (Participants) | 35
    Non-Boosted TDF Containing Regimens | 0.98 (1.44)
    Non TDF Containing Regimens: number analyzed (Participants) | 15
    Non TDF Containing Regimens | 1.02 (0.255)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: All enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
percentage of participants | 95.3 [89.3 to 98.5]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
percentage of participants | 1.9

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
percentage of participants
  SVR4 | 95.3 [89.3 to 98.5]
  SVR24 | 95.3 [89.3 to 98.5]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Time Frame: Up to 12 Weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
percentage of participants
  Week 1: number analyzed (Participants) | 105
  Week 1 | 25.7 [17.7 to 35.2]
  Week 2: number analyzed (Participants) | 103
  Week 2 | 68.0 [58.0 to 76.8]
  Week 4: number analyzed (Participants) | 103
  Week 4 | 92.2 [85.3 to 96.6]
  Week 6: number analyzed (Participants) | 103
  Week 6 | 99.0 [94.7 to 100.0]
  Week 8: number analyzed (Participants) | 102
  Week 8 | 100.0 [96.4 to 100.0]
  Week 10: number analyzed (Participants) | 102
  Week 10 | 100.0 [96.4 to 100.0]
  Week 12: number analyzed (Participants) | 102
  Week 12 | 100.0 [96.4 to 100.0]

5. Secondary Outcome: HCV RNA Change From Baseline/Day 1
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 101
  Change at Week 1 | -4.47 (0.606)
  Change at Week 2: number analyzed (Participants) | 101
  Change at Week 2 | -4.97 (0.577)
  Change at Week 4: number analyzed (Participants) | 102
  Change at Week 4 | -5.15 (0.560)
  Change at Week 6: number analyzed (Participants) | 103
  Change at Week 6 | -5.18 (0.572)
  Change at Week 8: number analyzed (Participants) | 102
  Change at Week 8 | -5.17 (0.575)
  Change at Week 10: number analyzed (Participants) | 102
  Change at Week 10 | -5.17 (0.575)
  Change at Week 12: number analyzed (Participants) | 102
  Change at Week 12 | -5.17 (0.575)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks
Number analyzed (Participants) | 106
percentage of participants | 1.9

7. Secondary Outcome: Percentage of Participants That Maintained HIV-1 RNA < 50 Copies/mL While On HCV Treatment
Time Frame: Up to 12 Weeks
Population: Participants in the Safety Analysis Set with available data were analyzed by TDF-containing ART at baseline:
  * Boosted TDF-containing regimens
  * Non-boosted TDF-containing regimens
  * Non TDF-containing regimens
Measure: Number; unit: percentage of participants
Groups:
- SOF/VEL 12 Weeks (Boosted TDF Containing Regimens): SOF/VEL (400/100 mg) FDC tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1. Data for participants who took boosted TDF-containing regimens (defined as regimens containing TDF and ritonavir (RTV) or cobicistat (COBI)-boosted protease inhibitors (PIs) or other agents (eg, elvitegravir (EVG)/COBI)) are summarized in this group.
- SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens): SOF/VEL (400/100 mg) FDC tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1. Data are summarized for participants who took non-boosted TDF-containing regimens (defined as regimens containing TDF and non-RTV or COBI-boosted PIs or other agents).
- SOF/VEL 12 Weeks (Non TDF Containing Regimens): SOF/VEL (400/100 mg) FDC tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1. Data are summarized for participants taking regimens that do not contain TDF.
Arm/Group | SOF/VEL 12 Weeks (Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non TDF Containing Regimens)
Number analyzed (Participants) | 56 | 35 | 15
percentage of participants
  Week 4: number analyzed (Participants) | 54 | 35 | 14
  Week 4 | 94.4 | 97.1 | 100
  Week 8: number analyzed (Participants) | 54 | 35 | 14
  Week 8 | 96.3 | 97.1 | 100
  Week 12: number analyzed (Participants) | 53 | 35 | 14
  Week 12 | 96.2 | 100 | 92.9

8. Secondary Outcome: Serum Creatinine Change From Baseline At the End of Treatment and At Posttreatment Week 12
Time Frame: Week 12; Posttreatment Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- SOF/VEL 12 Weeks (Boosted TDF Containing Regimens): SOF/VEL (400/100 mg) FDC tablet orally once daily in HCV treatment-naive and treatment-experienced (including treatment intolerant) participants with chronic HCV infection who were coinfected with HIV-1. Data for participants who took boosted TDF-containing regimens (defined as regimens containing TDF and RTV or COBI-boosted PIs or other agents (eg, EVG/COBI)) are summarized in this group.
Arm/Group | SOF/VEL 12 Weeks (Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non TDF Containing Regimens)
Number analyzed (Participants) | 56 | 35 | 15
mg/dL
  Change at Week 12: number analyzed (Participants) | 51 | 35 | 14
  Change at Week 12 | 0.09 (0.196) | 0.04 (0.107) | 0.00 (0.083)
  Change at Posttreatment Week 12: number analyzed (Participants) | 53 | 35 | 12
  Change at Posttreatment Week 12 | 0.04 (0.153) | 0.02 (0.142) | -0.06 (0.204)

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks Plus 30 Days
Description: Safety Analysis Set
Arm/Group | SOF/VEL 12 Weeks (Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens) | SOF/VEL 12 Weeks (Non TDF Containing Regimens)
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/35 | 0/15
Other Adverse Events (participants affected / at risk) | 34/56 | 19/35 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (Boosted TDF Containing Regimens) (N=56) | SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens) (N=35) | SOF/VEL 12 Weeks (Non TDF Containing Regimens) (N=15)
Localised infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (Boosted TDF Containing Regimens) (N=56) | SOF/VEL 12 Weeks (Non-Boosted TDF Containing Regimens) (N=35) | SOF/VEL 12 Weeks (Non TDF Containing Regimens) (N=15)
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Chest discomfort (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 16 | 7 | 3
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Headache (Nervous system disorders) | 7 | 6 | 1
Abnormal dreams (Psychiatric disorders) | 3 | 1 | 0
Depression (Psychiatric disorders) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years